CLINICAL TRIAL: NCT04747899
Title: Effects of Positional Release Technique for Myofascial Trigger Points of the Upper Trapezius With Forward Head Posture
Brief Title: Positional Release Technique for Myofascial Trigger Points of the Upper Trapezius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00865 Asad Ullah
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: myofascial trigger points of the upper trapezius; Positional Release technique; Neck Pain Disability index; Cranio vertebral angle
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Active Comparator): Traditional physical therapy ,Hot Pack, Muscle Stretching and Posture correction
  Interventions: Other: Traditional physical therapy
- Positional Release Technique (Experimental): Experimental group is given Positional Release Technique along with the hot pack, muscle stretching and posture correction.
  Interventions: Other: Positional release technique

INTERVENTIONS:
Other: Positional release technique — Experimental group is given Positional Release Technique along with the hot pack, muscle stretching and posture correction.
  Positional release technique position will maintained for almost 90 seconds. This technique will be repeated for three times each session, with 10 sec relaxation, 3 days/week.
  Upper trapezius stretching 5 repetitions×1 set, 3 days/ week. Total of 3 sessions were given each consisting of 30 min.
  Posture correction in ADLs as well as in working place by advising correct sitting posture, the participants will advised to relieve muscle tension after every 20-30 minutes of work by getting up; stretching the arm, shoulder, neck, and back muscles.
  Arms: Positional Release Technique
Other: Traditional physical therapy — Hot pack for 15-mins. Upper trapezius stretching 5 repetitions×1 set, 3 days/ week. Total of 3 sessions are given each consisting of 30 min.
  Posture correction in ADLs as well as in working place by advising correct sitting posture, the participants will advised to relieve muscle tension after every 20-30 minutes of work by getting up; stretching the arm, shoulder, neck, and back muscles.
  Arms: Traditional physical therapy

SUMMARY:
The aim of this research is to find the effects of Positional Release Technique (PRT) on pain, range of motion and neck disability index in patients with myofascial trigger points (MTRPs) of the upper trapezius with forward head posture (FHP). A Randomized control trial is conducted at Tehsil Head Quater (THQ) Civil hospital Wazirabad. The sample size is calculated through open epi tool is 32. The subjects are divided in two groups, 16 participants in experimental group and 16 in control group. The study duration is of six months. Sampling technique applied is purposive non probability sampling technique. Only 18-45 years participants with myofascial trigger points of the upper trapezius is included. Tools used in the study are Visual analog scale (VAS), Pain Pressure Threshold (PPT), active cervical contra-lateral flexion (ACLF), Cranio vertebral angle (CVA) and neck disability index (NDI). Data analyzed through Statistical Package for the Social Sciences (SPSS) version 23.

DETAILED DESCRIPTION:
Muscular and skeletal structures can change into an incorrect shape due to a reduction in physical activity and inappropriate posture habits in daily living. Kong YS et al defined Forward head posture (FHP) as a posture that adopts upper cervical extension and lower cervical flexion. The center of gravity of the head in this posture is positioned at the front rather than the vertebral body weight.

FHP weakens the deep cervical flexor muscle, the mid thoracic rhomboid muscle for scapular retraction, and the mid and lower trapezius muscles. FHP also shortens the pectoralis major and neck extension muscles. Upper trapezius muscle activity is increased more in FHP than in correct anatomic positions, and most patients complain of pain from muscle overuse.

The craniovertebral angle (CVA) is defined as an angle made by the intersection of a line joining the midpoint of the tragus of ear to the skin overlying the C7 spinous process and a horizontal line passing through the C7 spinous process. There is a correlation between FHP, neck pain, and CVA. One of the studies reported that subjects having smaller CVA had FHP and were prone to have increased severity of neck pain.

D'souza CJ et al stated that positional Release Therapy (PRT) is a noninvasive treatment which can be used in conjunction with several electrical modalities. In this technique, in order to facilitate restoration of normal tissue length and to treat excessive muscle tension or spasm, tissues are placed in a Position of comfort for a brief period (90 sec) to resolve the associated dysfunction.

In 2017 a study conducted which shows that PRT has beneficial effects on myofascial trigger points (MTrPs). In this regard, Kelencz et al. reported that PRT is effective in reducing pain and muscle tension among patients with upper-trapezius MTrPs. Amini A et al studied on 30 female university students, who were identified with latent MTrPs of the upper trapezius, according to the results, both Manual Passive Muscle Shortening (MPMS) and PRT were effective techniques in immediate pain relief of upper-trapezius MTrPs.

Kojidi MM et al concluded that Positional Release Therapy was found to be effective in reducing pain and increasing Pressure pain threshold in three treatment sessions in 19-45 year-old female computer users with at least 2 h of work and with latent upper trapezius trigger points. Mohamadi M et al state that PRT is a potential treatment option with no reported side effects for patients with Tension Type Headache (TTH).

In general, PRT and Therapeutic Massage were both successful at decreasing MTrP sensitivity and stiffness. However, there appeared to be a slight benefit for pain reduction with PRT up to 2 days post treatment.

Varshney K et al concluded that the patients who received positional release therapy along with moist heat pack has more impact on pain and disability as compared to those received deep transverse friction massage along with moist heat pack follow-up 4 weeks protocol.

Study concluded that the difference from 1st to 21th day in VAS &NDI score which shows that Positional release therapy (PRT) is more effective than conventional Physiotherapeutic intervention in order to decrease pain and disability in patients with no-specific neck pain.

Manzoor S et al treated a 62 year female who was suffering tension type headache from last 14 months was treated by combined positional release therapy and ischemic compression in 6 sessions, concluded that combination of positional stretch and Ischemic compression is effective treatment for patients with trigger points in cervical muscles, most commonly upper trapezius and sternocleidomastoid causing cervicogenic headache.

There is poor evidence regarding the effects of PRT on MTRPs with forward head posture on Cranio-vertebral angle. So this study aims to find the effectiveness of PRT for myofascial trigger points of the upper trapezius with forward head posture as there is less literature available about the gender based effect of PRT, as most of the studies have done on female population, basically this study will target the effect of PRT on male computer users with FHP on Pain, ROM, disability and Cranio vertebral angle.

ELIGIBILITY:
Inclusion Criteria:

* Pain intensity of at least 3 on VAS.
* Presence of palpable taut band & at least one active trigger point in upper trapezius. Diagnosis of trigger point will confirm by following criteria given by Travel & Simon.
* CVA less than 50 degrees while standing.
* At least 6 hours in sitting position and work via computers per day

Exclusion Criteria:

* Diagnosis of fibromyalgia & RA.
* Diagnosis of cervical Radiculopathy or Myelopathy
* History of a whiplash injury
* History of cervical spine and shoulder surgery
* Having undergone Trigger point therapy within the past month prior to the study
* Drug intake (anti-inflammatory medication during treatment sessions)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — computer users ' Male with Forward head posture due to upper trapezius Triggers point at least one taut band
Enrollment: 32 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 12th day
  Changes from base line Northwick disability index was developed first in Northwick Park hospital, England. It was designed to measure the neck pain and disability over time. It consists of 10, five parts sections. At the end, score is calculated by dividing the obtained score by total (50) multiplied by 100. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'.

SECONDARY OUTCOMES:
Visual analog scale | 12th day
  Changes from base Line Visual Analog Scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
ROM Active Contra Lateral Flexion (ACLF) | 12th day
  Changes from the Baseline ROM range of Motion of Active Contra Lateral Flexion (ACLF) is taken with the Help of Goniometry. Subjects sit upright and laterally flex their head towards the opposite side of involvement and the motion was stopped once the available ROM was completed.
Pain Pressure Threshold (PPT | 12th day
  Changes from the Baseline Pain Pressure Threshold (PPT) was taken with the Help of Algometer.
Cranio vertebral angle (CVA) | 12th day
  Changes from the baseline Cranio vertebral angle is measured by intersection of a horizontal line passing through the C7 spinous process and a line joining the midpoint of the tragus of the ear to the skin overlying the C7 spinous process.

CONTACTS AND LOCATIONS:
Overall Officials: Saira Waqqar, PHD*, Principal Investigator — Riphah International University
Locations (1):
- THQ Civil Hospital, Wazirabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee DY, Nam CW, Sung YB, Kim K, Lee HY. Changes in rounded shoulder posture and forward head posture according to exercise methods. J Phys Ther Sci. 2017 Oct;29(10):1824-1827. doi: 10.1589/jpts.29.1824. Epub 2017 Oct 21. PMID 29184298
- [Background] Kong YS, Kim YM, Shim JM. The effect of modified cervical exercise on smartphone users with forward head posture. J Phys Ther Sci. 2017 Feb;29(2):328-331. doi: 10.1589/jpts.29.328. Epub 2017 Feb 24. PMID 28265167
- [Background] Kim SY, Koo SJ. Effect of duration of smartphone use on muscle fatigue and pain caused by forward head posture in adults. J Phys Ther Sci. 2016 Jun;28(6):1669-72. doi: 10.1589/jpts.28.1669. Epub 2016 Jun 28. PMID 27390391
- [Background] Sikka I, Chawla C, Seth S, Alghadir AH, Khan M. Effects of Deep Cervical Flexor Training on Forward Head Posture, Neck Pain, and Functional Status in Adolescents Using Computer Regularly. Biomed Res Int. 2020 Oct 5;2020:8327565. doi: 10.1155/2020/8327565. eCollection 2020. PMID 33083487
- [Background] Mohammadi Kojidi M, Okhovatian F, Rahimi A, Baghban AA, Azimi H. The influence of Positional Release Therapy on the myofascial trigger points of the upper trapezius muscle in computer users. J Bodyw Mov Ther. 2016 Oct;20(4):767-773. doi: 10.1016/j.jbmt.2016.04.006. Epub 2016 Apr 7. PMID 27814857
- [Background] Amini A, Goljaryan S, Shakouri SK, Mohammadimajd E. The Effects of Manual Passive Muscle Shortening and Positional Release Therapy on Latent Myofascial Trigger Points of the Upper Trapezius: A Double-Blind Randomized Clinical Trial. Iranian Red Crescent Medical Journal. 2017 Sep;19(9).
- [Background] Varshney K, Raghav S, Singh A. A study to compare the effect of positional release technique (PRT) versus deep transverse friction massage (DTFM) on pain and disability in patients with mechanical neck pain.
- [Background] Varshney K, Raghav S, Singh A, Meena R K, Sharma S. Short term effect of Positional Release Therapy versus conventional Physiotherapeutic programme on pain and disability among undergraduate Physiotherapy students with nonspecific neck pain: A Pilot Study. Subharti J of Interdisciplinary Research, April 2019; Vol. 2: Issue 1, 7-11.
- [Background] Manzoor S, Afzal F. Effect of Combined positional stretch and ischemic compression on Cervicogenic Headache. Headache.;1:2.